CLINICAL TRIAL: NCT01051271
Title: Prophylaxis Against Metoclopramide-Induced Akathisia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PAU-200/1563
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-07

CONDITIONS: Akathisia
Keywords: metoclopramide; akathisia; midazolam; diphenhydramine; metoclopramide induced akathisia
MeSH Terms: conditions — Psychomotor Agitation | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- diphenhydramine (Active Comparator)
  Interventions: Drug: midazolam
- saline (Placebo Comparator)
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: midazolam — midazolam 1.5 mg

SUMMARY:
ABSTRACT

Study Objective:

To compare the effects of midazolam and diphenhydramine for the prevention of metoclopramide induced akathisia.

Methods:

This randomized, double-blind and controlled trial aimed to investigate co-administered midazolam versus diphenhydramine in the prophylaxis of metoclopramide induced akathisia. Patients 18 through 65 years of age who presented to the ED with primary or secondary complaints of nausea and/or moderate to severe vascular type headache were eligible for this study. Patients were randomized to one of the fallowing three groups: (1) metoclopramide 10 mg + midazolam 1.5 mg (2) metoclopramide 10 mg + diphenhydramine 20 mg (3) metoclopramide 10 mg + placebo. Metoclopramide was administered as a 2 minutes bolus infusion. Midazolam, diphenhydramine and normal saline solution administered as a 15 minutes slow infusion. Whole procedure was observed, akathisia and sedation scores and vital changes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 through 65 years of age and 50-90 kg of weight who presented to the ED with primary or secondary complaints of nausea and/or moderate to severe vascular type headache were eligible for this study.

Exclusion Criteria:

* Patients who had liver and renal insufficiency
* Electrolyte imbalance
* Acute respiratory symptoms
* Chronic obstructive pulmonary disease
* Blood pressure less than 90/60 mmHg
* Uncooperative individuals
* Pregnant or lactating
* Pre-existing motor disorder
* Restless legs syndrome-parkinson's disease
* Organic brain disorder, (dementia etc.), epilepsy
* Admitted to the ED due to acute psychiatric symptoms
* Deprived mental status
* Advanced hearing loss
* Malnutrition
* Acute asthma attack
* Serious physical illness, especially glaucoma, prostatic hypertrophy, or cardiac disease
* Had a contraindication to anticholinergic medications
* Within 3 days of study entry patients who had taken an antiemetic antihistaminic, antipsychotic, antispasmodic, alpha-blocker, or Ca++2-channel blocker, or within 2 weeks of study entry patients who had taken an antidepressant, barbiturate, benzodiazepine, other sedative/hypnotic, opioid, lithium, or illicit sympathomimetic agent were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
akathisia and sedation scores